CLINICAL TRIAL: NCT00172913
Title: National Taiwan University Hospital
Brief Title: Aberration-Free Refraction Correction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700324
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Myopia
Keywords: Wavefront Aberration; LASIK; Contrast Sensitivity; Visual Performance; Ablation Profile
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
In the interest of improving visual quality after LASIK we have designed a multifaceted study to test the theoretical, physical, biomechanical and functional effects of commercial and independently designed aspherical ablation profiles.

DETAILED DESCRIPTION:
The quality of an image on the retina is determined by the optical system of the eyeball, which is dominated by the refractive contribution of the optically powerful cornea. The large difference in refractive index between air and the cornea is the basis for anterior corneal refractive surgery such as Laser in situ Keratomileusis (LASIK) which reshapes the naturally aspherical cornea to correct a patient's vision. In addition to correcting refractive errors, current spherical LASIK treatments have been shown to increase ocular wavefront aberrations which can reduce visual quality postoperatively. Modifications of the corneal-ablation algorithm have been suggested to correct this issue.

Until recently, most ablation algorithms have relied on the Munnerlyn formula, which assumes the anterior corneal surface to be spherical before and after refractive surgery. One concept for customized ablation is to apply an ablation during the surgical procedure which has been adapted to the patient's own aberration pattern. Since custom ablation algorithms are proprietary and we do not know how they consider the role of asphericity.

Precisely altering the corneal asphericity after refraction surgery is a complex phenomenon which includes biomechanical effects. Thus, knowledge of the cornea's response to the different aspherical ablation profiles is vital for understanding corneal properties and prediction of surgical outcomes.

This study will involve computer simulation of ablation profiles for the respective lasers, interferometric analysis of actual ablation profiles on PMMA plates, optimization for visual correction, functional studies of the short and long term effects of the profiles on in vivo human corneas, and quantitative subjective (questionnaire and visual tests) and objective analysis (calculation of retinal image quality metrics) and comparison of the effects aspherical ablation profiles on visual quality. The completion of the project will lead to objective evaluation of current ablation profiles as well as the development and evaluation of new optimized laser refractive surgery procedures with improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* This will be a prospective study including at least 60 patients. The initial study group will include 6-10 patients. Both eyes of enrolled patients should be included in the study unless exclusion criteria prevent it. The primary efficacy variables for this study are wavefront error, visual acuity, autorefraction and contrast sensitivity. Subjects will be followed over a 3 month period. A proposed examination schedule is listed in Table 1.

Eyes will also be divided into groups by refractive error: Low myopia 0-3D, moderate myopia 3-6D, and high myopia 6-9 D and very high myopia > 9D MSRE. The size of the Optical Zone and Transitional Zone is measured, and results are compared for patients of similar refractive error (+/- 0.5 S +/- 0.5 C). Analysis is carried out using a matrix analysis of the total refractive error, comparison of Visual Acuity, Contrast Sensitivity and Responses on a Questionnaire to assess the patient's quality of vision.

Equal numbers of eyes from each of the four refractive error groups and from each of the three treatment groups (OATZ profile 5, OATZ profile 6, conventional) will be measured.

We will consider patients operated on by the same doctor (Dr. Lin). We will also compare treatments of patients and wavefront maps of patients who have similar spherical and cylindrical refractive errors.

Table 1. Examination Schedule (Definitions) Visit Time Preoperative Within 30 days of surgery Operative Day Day of surgery

1 Month postop 3-5 weeks following surgery 3 Months postop 10-14 weeks following surgery

Exclusion Criteria:

* Patients will be excluded if they have a history of ocular pathology, previous ocular surgery, thin corneas (preoperatively calculated minimal residual bed < 250um) or fit into the group of the usual exclusionary criteria (e.g. irregular astigmatism, asymmetric astigmatism, unstable refraction).

Possible additional exclusion criteria include no previous refractive surgery, no hyperopia, preop BSCVA 20/25 or better, ages from 21-60 years old, astigmatism above 2D, difficult cases and equal numbers of men and women

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06; Study Completion 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, MD,PHD, Principal Investigator — National Taiwan University Hospiyal
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan